CLINICAL TRIAL: NCT06230614
Title: Effect of Diluent Volume on Colistin Inhalation Therapy for Mechanically Ventilated Respiratory Patients
Brief Title: Effect of Diluent Volume on Colistin Inhalation Therapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fu Jen Catholic University (Other)
Responsible Party: Principal Investigator, Ke-Yun, Chao, Group leader of Respiratory Therapists, Fu Jen Catholic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: FJUH112294
Record Dates: First submitted 2024-01-21; First posted 2024-01-30 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Inhalation Pneumonia
Keywords: Colistin; antibiotic; inhalation therapy; diluent volume; randomized controlled trial
MeSH Terms: conditions — Pneumonia, Aspiration | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Colistin 1 MU in normal saline 1 ml (Active Comparator): 1 MU of colistin in a total volume of 6 ml, diluted with a 1:1 ratio in normal saline (0.9%)
  Interventions: Other: Colistin 1 MU in normal saline 1 ml
- Colistin 1 MU in normal saline 2 ml (Experimental): 1 MU of colistin in a total volume of 12 ml, diluted with a 1:2 ratio in normal saline (0.9%)
  Interventions: Other: Colistin 1 MU in normal saline 2 ml

INTERVENTIONS:
Other: Colistin 1 MU in normal saline 1 ml — Colistin 1 MU diluted in normal saline 1 ml, total volume of 12 ml
  Arms: Colistin 1 MU in normal saline 1 ml
Other: Colistin 1 MU in normal saline 2 ml — Colistin 1 MU diluted in normal saline 2 ml, total volume of 12 ml
  Arms: Colistin 1 MU in normal saline 2 ml

SUMMARY:
The aim of this study is to investigate the impact of different diluent volumes for the same dosage of colistin in mechanically ventilated respiratory patients receiving colistin inhalation therapy. The study aims to determine whether the diluent volume has an effect on clinical outcomes, including ICU length of stay, total hospitalization duration, duration of respiratory support within 28 days, mortality rates within 28 days and 90 days, as well as analyze the pharmacokinetic profile of colistin in blood and bronchoalveolar lavage fluid. Additionally, the study will evaluate the incidence of nebulizer malfunctions and blockages. The findings of this research will help identify the optimal diluent volume for colistin inhalation therapy in clinical practice.

DETAILED DESCRIPTION:
Background： Colistin is an antibiotic used to treat infections caused by multidrug-resistant Gram-negative bacteria. In recent years, it has been widely utilized as an inhaled antibiotic for the treatment of respiratory infections in critically ill patients on mechanical ventilation. Despite the increasing use of colistin inhalation therapy for ventilator-associated pneumonia, the clinical impact of diluent volume on nebulization efficiency remains unclear.

Study Design： A single-center, prospective, randomized controlled trial.

Methods： The study plans to enroll 60 participants. Colistin inhalation therapy will be administered using a blocked stratified random allocation. The control group will receive colistin 6 MU diluted in 6 ml of normal saline (1 MU per 1 ml), while the experimental group will receive colistin 6 MU diluted in 12 ml of normal saline (1 MU per 2 ml). The dosage, frequency, and administration method of colistin inhalation will follow the clinical standard of 6 MU, administered every 8 hours, continuously for 7 days.

Effect： The investigators anticipate that the clinical outcomes and pharmacokinetics of colistin inhalation therapy will not differ significantly between different diluent volumes. Based on comprehensive evaluation, a diluent volume of 12 ml is considered more suitable than 6 ml for the dilution of colistin.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to the Intensive Care Unit.
* Age greater than 18 years and using a ventilator due to acute respiratory failure.
* Requires inhalation colistin treatment as determined by the disease.
* Sign the written informed consent form.

Exclusion Criteria:

* Renal failure requiring renal dialysis.
* Receiving both inhaled colistin and intravenous colistin treatments.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-03-10 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Drug concentration | One hour post inhalation therapy with colistin on the third day of treatment
  Drug concentration in bronchoalveolar lavage fluid and blood

CONTACTS AND LOCATIONS:
Overall Officials: Ke-Yun Chao, PhD, Principal Investigator — Fu Jen Catholic University Hospital
Locations (1):
- Fu Jen Catholic University Hospital, Fu Jen Catholic University, New Taipei City, Taiwan